CLINICAL TRIAL: NCT02885467
Title: Saphenous Nerve Brach Burial for Preventing Neuralgia After Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Nerve Burial for Preventing Neuralgia After Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by IRB
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB 2013-281
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Neuralgia; Osteoarthritis of the Knee
Keywords: Total Knee Arthroplasty
MeSH Terms: conditions — Neuralgia; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Standard total knee arthroplasty performed through medial parapatellar approach
  Interventions: Procedure: Standard total knee arthroplasty
- Intervention (Experimental): Total knee arthroplasty performed through medial parapatellar approach with identification, ligation, and burial of saphenous nerve branches
  Interventions: Procedure: Total knee arthroplasty with Saphenous nerve burial

INTERVENTIONS:
Procedure: Total knee arthroplasty with Saphenous nerve burial
  Arms: Intervention
Procedure: Standard total knee arthroplasty
  Arms: Control

SUMMARY:
This is a randomized study investigating whether identification, ligation, and burial of superficial branches of the saphenous nerve crossing the surgical field during total knee arthroplasty reduces the rate of post-operative anterior knee pain and neuralgia compared to standard total knee arthroplasty.

DETAILED DESCRIPTION:
Anterior knee pain is common after total knee arthroplasty. The incision necessarily travels through the path of a cutaneous nerve - branches of the saphenous nerve. Historically, no effort has been made to separate these branches and bury them away from the surgical scar. It has been noted that some patients develop a painful neuroma, that once resected results in a pain free knee. Investigators are trying to study if identification, ligation, and proper burial of the nerve can prevent the development of neuralgia compared to the typical surgical approach which ignores the nerve branches completely.

ELIGIBILITY:
Inclusion Criteria:

* Must have symptomatic knee osteoarthritis under consideration for total knee arthroplasty
* Must be willing to undergo randomization

Exclusion Criteria:

* Age <18 or >80 years
* Known pre-operative diagnosis of neuralgia, complex regional pain syndrome, or neuropathy, about the operative lower extremity
* Known pre-operative psychiatric disorder requiring medication
* Previous surgery about the operative knee
* BMI > 40 kg/m2 (potential increased risk of soft tissue dissection through adipose)
* Ongoing pre-operative narcotic use in excess of 20 mg morphine equivalents per day for at least one month or pre-operative intravenous drug use (increased potential for complex regional pain syndrome and neuralgia, increased likelihood to require greater post-operative analgesia)
* Ongoing pre-operative use of neuropathic pain medications (gabapentin, pregabalin, amitriptyline, etc.)
* Medical comorbidities (American Society of Anesthesiologists grade > 3 or deemed unfit by consulting internist) precluding elective TKA
* Significant language barrier (reading comprehension less than 8th grade reading level) or mental condition precluding accurate self-assessment of knee pain or function.
* Severe medication allergies to permissible post-operative analgesics (acetaminophen, tramadol, oxycodone, oxycontin, dilaudid)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Incidence of neuralgia | 2 years
  Measured by DN4 validated scoring tool

SECONDARY OUTCOMES:
Oxford Knee Score | 2 years
Kneeling weight | 2 years
  Ability to kneel with body weight on affected knee

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Union Memorial Hospital, Baltimore, Maryland, United States